CLINICAL TRIAL: NCT04982055
Title: Intravenous Versus Subcutaneous Administration of Low Molecular Weight Heparin for Thromboprophylaxis in Critically Ill Patients: a Randomized Controlled Trial
Brief Title: Intravenous Versus Subcutaneous Administration of Low Molecular Weight Heparin for Thromboprophylaxis in Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinique Saint Pierre Ottignies (Other)
Responsible Party: Principal Investigator, Nicolas De Schryver, Principal investigator, Clinique Saint Pierre Ottignies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IV vs SC LMWH ICU
Record Dates: First submitted 2021-07-08; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Nadroparin; Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous group (Experimental)
  Interventions: Drug: Nadroparin (intravenous Infusion)
- Subcutaneous group (Active Comparator)
  Interventions: Drug: Nadroparin (subcutaneous group)

INTERVENTIONS:
Drug: Nadroparin (intravenous Infusion) — Intravenous route of administration over a 4-hours infusion of nadroparin 3800 IU
  Arms: Intravenous group
Drug: Nadroparin (subcutaneous group) — Subcutaneous route of administration of nadroparin 3800 IU
  Arms: Subcutaneous group

SUMMARY:
Objective: To compare the pharmacokinetic profiles of intravenous versus subcutaneous route of administration of LMWH for thromboprophylaxis in critically ill patients

DETAILED DESCRIPTION:
The study is a prospective, monocentric, randomized trial. Patients are randomized to the IV route of administration over a 4-hours infusion of nadroparin 3800 IU or to the SC route of administration. Randomization is stratified according to the need for vasopressor or not. Anti-Xa activity is measured at baseline, and at 1, 2, 4, 6, 8, 12 and 24 hours after the administration was started.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients > 18 years old admitted in the ICU, and for whom thromboprophylaxis is indicated

Exclusion Criteria:

* renal failure determined by glomerular filtration rate (GFR) < 30 ml/min or need for renal replacement therapy
* liver cirrhosis
* intravascular disseminated coagulation
* contra-indication to thromboprophylaxis for any reason as decided by the treating physician, or indication for therapeutic dosing anticoagulation (recent thrombo-embolic event, atrial fibrillation,…)
* patients receiving low dose of vasopressor (norepinephrine < 0.25 mcg/kg/min) to allow stratification and comparison between patients not on vasopressors and patients with a significant dose of vasopressors (norepinephrine ≥ 0.25 mcg/kg/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Peak anti-Xa activity | Peak anti-Xa activity obtained 4 hours after start of low molecular weight heparin administration
  Peak anti-Xa activity obtained 4 hours after start of low molecular weight heparin administration

SECONDARY OUTCOMES:
Trough anti-Xa activity | Trough anti-Xa activity measured 24 hours after start of low molecular weight administration
  Trough anti-Xa activity measured 24 hours after start of low molecular weight administration
AUC (0-24h) | 0-24 hours
  Area under the curve 0-24 hours of anti-Xa activity after start of low molecular weight heparin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Schryver N, Serck N, Eeckhoudt S, Laterre PF, Wittebole X, Gerard L. Pharmacokinetic profiles of intravenous versus subcutaneous administration of low molecular weight heparin for thromboprophylaxis in critically ill patients: A randomized controlled trial. J Crit Care. 2022 Aug;70:154029. doi: 10.1016/j.jcrc.2022.154029. Epub 2022 Apr 2. PMID 35381407